CLINICAL TRIAL: NCT06026293
Title: Retrospective and Prospective Study Aimed At the Pharmacoeconomic Evaluation of the Cost/effectiveness Ratio of Physical Exercise on the Prognosis of Non-alcoholic Fatty Liver Disease (NAFLD)
Brief Title: Pharmacoeconomic Evaluation of the Cost/effectiveness Ratio of Physical Exercise on Non-alcoholic Fatty Liver Disease
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Collaborators: Antonella Bianco (Unknown); Pietro Trisolini (Unknown); Giuseppe Dalfino (Unknown)
Responsible Party: Principal Investigator, Maurizio Gaetano Polignano, principal investigator, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Other Study IDs: CER_study
Record Dates: First submitted 2023-08-30; First posted 2023-09-07 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: Non-alcoholic fatty liver desease; Cost/effectivness; Physical activity
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- subjects that participates to a previous clinical trial

SUMMARY:
Physical inactivity and poor dietary habits are associated with an increased risk of obesity and chronic disease (World Health Organization, 2019; Glanz and Bishop, 2010). Conversely, higher levels of total physical activity result in a reduced risk of cardiovascular disease, breast and colon cancer, and diabetes (Kyu et al., 2016). Similarly, consumption of the minimum recommended level (600 g per day) of fruit and vegetables is associated with a lower risk of cardiovascular disease and cancer (Ezzati et al., 2004). However, despite these recognized benefits, unhealthy diet and physical inactivity are still major contributors to poor health and rising health care costs. Worldwide, physical inactivity accounted for 13.4 million disability-adjusted life years (DALYs) in 2013 and cost $53.8 billion to health systems and an additional $13.7 billion in productivity due to deaths attributable to physical inactivity (Ding et al., 2016).

Pharmacoeconomics, or the economic evaluation of treatments aimed at maintaining the health of the population, is a set of evaluation models used to identify the value (convenience) and the overall economic impact of a possible treatment.

The results of economic evaluations help decision makers inform their choice. Their advantage is that the result is obtained by applying known and validated models, and everyone can know the basis of the decision (evidence-based decision making). The clinical-economic value and the overall financial impact must be compared with the willingness to pay the related costs.

Economic evaluations are a tool for defining the value of a medicine in terms of cost-opportunity, from the point of view of the patient, the NHS and society as a whole.

The definition of "value" is very broad, multidimensional and includes concepts from many disciplines, beyond economics. Specifically, economic evaluations that take into consideration new medicines, innovative or not, the value is given by the marginal utility that the patient, the NHS and/or society can obtain from its acquisition. In this regard, the measurement of years of life gained in full quality of life (QALY - quality-adjusted life years) is widely applied to medicines in various regulatory contexts, albeit with the awareness that it is not able to capture all the elements that contribute to value (Carletto, A et al.; Drummond, M. F)

ELIGIBILITY:
Inclusion Criteria:

* Being affected by NAFLD in the observation period (2018-2020)
* Participating in health promotion activities by performing physical exercise under the supervision of the institution's kinesiologists

Exclusion Criteria:

* Patient deceased
* Patient who does not agree to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population was affected by NAFLD in the observation period (2018-2020), participating in health promotion activities by performing physical exercise under the supervision of the institution's kinesiologists
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
Cost/effectiveness Ratio | 3 years
  to define the economic value in terms of CER (Cost/Effectiveness Ratio) and ICER (Incremental Cost/Effectivness Ratio) of physical exercise in the treatment of NAFLD in patients who already have comorbidities for metabolic/cardiometabolic diseases.

SECONDARY OUTCOMES:
long term foresight of an healthy policy | 3 years
  identify the potential savings in terms of costs (direct and indirect) of physical exercise on patients suffering from NAFLD through the use of a predictive scenario developed through the use of the MAFEIP (Monitoring and Assessment Framework for the European Innovation Partnership on Active and Healthy Aging).

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Gaetano Polignano, Principal Investigator — IRCCS "Saverio de Bellis"
Locations (1):
- Irccs Saverio de Bellis, Castellana Grotte, Bari, Italy

REFERENCES:
- [Derived] Polignano M, Bianco A, Guido D, Trisolini P, Franco I, Bonfiglio C, Giannelli G. Economic value and clinical association of a supervised lifestyle-improving program for MASLD. Front Pharmacol. 2026 Jan 16;16:1708451. doi: 10.3389/fphar.2025.1708451. eCollection 2025. PMID 41625336